CLINICAL TRIAL: NCT04484194
Title: Assessing Health Electronically for Adolescent and Young Adult Oncology (AHEAD)
Brief Title: Assessing Health Electronically for Adolescent and Young Adult Oncology
Acronym: AHEAD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Collaborators: Tickit Health Solutions (Unknown)
Responsible Party: Principal Investigator, Tyler Ketterl, MD, MS, Assistant Professor, Department of Pediatrics, Seattle Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: STUDY00002661
Record Dates: First submitted 2020-07-14; First posted 2020-07-23 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Risk Reduction Behavior
MeSH Terms: conditions — Risk Reduction Behavior

STUDY DESIGN:
Intervention Model Description: Single center pilot feasibility study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- eHA Screening (Experimental): Patients receiving eHA screening tool.
  Interventions: Behavioral: Check Yourself - Oncology

INTERVENTIONS:
Behavioral: Check Yourself - Oncology — A validated AYA-targeted electronic health assessment (eHA) screening tool for use in oncology clinics.
  Other Names: Electronic Health Assessment (eHA)

SUMMARY:
The purpose of this study is to modify an existing Seattle Children's Hospital investigator-developed, patient-centered, electronic health assessment (eHA) called "Check Yourself" for AYAs with cancer. The investigators will then evaluate the new eHA prototype for feasibility and acceptability among AYAs with cancer and their oncology providers.

DETAILED DESCRIPTION:
Unmet needs among Adolescents and Young Adults (AYAs) with cancer translate to poor physical and psychosocial outcomes. This is particularly true when it comes to AYA sexual health. Our team has found that intimate relationships and risky health behaviors are common among AYAs during their cancer experience, that oncology clinicians rarely ask about these behaviors, and that AYAs rarely volunteer to share these behaviors. As a result, AYAs with cancer are deprived of the surveillance, anticipatory guidance, and normative support participants would have received if participants were well. Currently there is no standard screening process for risk behaviors and the recommended psychosocial screening for AYAs in the SCH oncology clinic setting. To address this problem, the investigators propose to adapt a validated AYA-targeted electronic health assessment (eHA) screening tool for use in oncology clinics.

The purpose of this study is to modify an existing Seattle Children's Hospital investigator-developed, patient-centered, electronic health assessment (eHA) for AYAs with cancer. The investigators will then evaluate the new eHA prototype for feasibility and acceptability among AYAs with cancer and their oncology providers.

AIM 1. To evaluate the modified eHA program prototype for feasibility, acceptability, and process measures. The investigators will enroll a cohort of N=25 AYAs with cancer and N=10 providers from our institution to "beta-test" the program.

Hypothesis 1: There will be applicable and nonapplicable eHA content for AYAs with cancer in the current electronic health assessment (eHA) tool in addition to content relative to AYAs with cancer that should be developed and added.

Hypothesis 2: AYAs will report that the modified AYA oncology specific eHA is both useful and easy to use. Additionally, oncology providers will report that the eHA tool was useful and positively impacted patient care.

ELIGIBILITY:
Inclusion Criteria:

* Eligible adolescents and young adults will be 13 to 29 years old, have an oncologic diagnosis for which they are receiving cancer directed therapy, have an appointment to see an SCH oncology provider and will be able to understand English.
* Eligible oncology providers will either be a Physician (Fellow or Attending) or Advance Practice Provider (Nurse Practitioner or Physicians Assistant), have an appointment to see an adolescent or young adult receiving cancer directed therapy receiving who is also enrolled on the study.

Exclusion Criteria:

* Participants will be excluded from the study if they do not meet age requirements, do not have an appointment in oncology clinic, lack the means to complete follow-up interviews (i.e., has neither telephone nor internet access), and/or are not able to understand English. Our experience in the Seattle region is that, because of English Language Learning schooling supports, inability to read or understand English is a barrier for <0.5% of adolescents. Thus, we do not anticipate that language restrictions will significantly limit the demographic distribution of our participants.

Ages: 13 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Actual)
Dates: Start 2021-04-15 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Determine the feasibility of eHA tool in AYA patients undergoing cancer directed therapy. | 12 months
  Determine the feasibility of Electronic Health Assessment (eHA) tool in AYA population with cancer diagnosis using the feasibility of intervention measure (FIM) tool survey.
Determine the acceptability of eHA tool in AYA patients undergoing cancer directed therapy. | 12 months
  Determine the acceptability of Electronic Health Assessment (eHA) tool in AYA population with cancer diagnosis using the acceptability of intervention measure (AIM) tool survey.
Determine the usability of eHA tool in AYA patients undergoing cancer directed therapy. | 12 months
  Determine the usability of Electronic Health Assessment (eHA) tool in AYA population with cancer diagnosis using the usability of intervention of appropriateness measure (IAM) tool survey.

CONTACTS AND LOCATIONS:
Overall Officials: Tyler G Ketterl, MD, MS, Principal Investigator — Seattle Children's Hospital
Locations (1):
- Seattle Children's, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No